CLINICAL TRIAL: NCT00366197
Title: Prediction of Weaning Outcomes by Using Rate of Change of Rapid Shallow Breathing Index
Status: Terminated | Type: Observational
Sponsor: Atlantic Health System (Other)
Other Study IDs: Rapid Shallow Breathing Index
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Rapid Shallow Breathing
Keywords: Rapid Shallow Breathing Index; Mechanical Ventilation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This trial examines weaning outcomes using the rapid shallow breathing index rate.

DETAILED DESCRIPTION:
We hypothesize that the trend of the Rapid Shallow Breathing Index or RSBI rate, is a better predictor of weaning outcome than the RSBI as a single value during the weaning trial. patients are recruited during a weaning trial on t-piece and the RSBI during what the RSBI is measured periodically. The outcome is ventilatory status at 24 hours after the weaning trial.

ELIGIBILITY:
Inclusion Criteria:

* Requires need of mechanical ventilation for > 48 hours with a tube size no smaller than 7.5

Exclusion Criteria:

* Healthy volunteers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and Female
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-01; Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Fiel, MD, Principal Investigator — Atlantic Health System; Harris Rana, MD, Principal Investigator — Atlantic Health System; Salvatore Ruggiero, MD, Principal Investigator — Atlantic Health System; Erwin Oei, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Morristown Memorial Hospital, Morristown, New Jersey, United States